Statistical analysis for the Cytarabine (Ara-C) in Children With Acute

Promyelocytic Leukemia (APL) (NCT01191541)

## **Principal Investigator**

## Xiaofan Zhu MD

<sup>1</sup>Department of Pediatrics, State Key Laboratory of Experimental Hematology and Division of Pediatric Blood Diseases Center, Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China.

## Statistical analysis

The primary objective was to demonstrate the noninferiority of DNR alone compared to DNR+Ara-C in terms of the DFS rate at 2 years. Assuming a 95% rate of DFS in the two groups, a margin of -14%, 5% type 1 error, and 80% power, 31 evaluable patients per group were required to draw a noninferiority conclusion.

The characteristics of all of the included patients were summarized using cross-tabulations (for categorical variables) and quantiles (e.g., the median; for continuous variables). Nonparametric tests were used to analyse comparisons between groups (i.e.,  $\chi^2$  and Fisher's exact tests for categorical variables). EFS, DFS and OS were estimated using the Kaplan -Meier method, and log-rank tests were used for comparisons. All P values were two-sided, and those with values of 0.05 or less were considered to be statistically significant. All statistical analyses were performed using SPSS software.